CLINICAL TRIAL: NCT02171936
Title: Chronic Pain and Social Vulnerability: Prevalence and Predictive Factors of the Social Vulnerability in Evaluation and Treatment of the Pain Center (CETD)
Acronym: PRECAPAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0194
Record Dates: First submitted 2014-06-16; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Pain
Keywords: Pain; Precariousness; EPICES Score; CETD
MeSH Terms: conditions — Chronic Pain; Pain

GROUPS / COHORTS (1):
- chronic pain
  Interventions: Other: Questionnaire EPICES (Evaluation of the Precariousness and the Disparities of Health for the Centers of Examination of Health).

INTERVENTIONS:
Other: Questionnaire EPICES (Evaluation of the Precariousness and the Disparities of Health for the Centers of Examination of Health).

SUMMARY:
In the care of the chronic pain in pain's department, pain consultation or Evaluation and Treatment of the Pain Center (CETD), the patients are often in a situation of physical and psychic suffering which requires a multidisciplinary follow-up. So, 19 percent of the chronic painful patients lost their employment, are "disintegrated" because of their pain, this being able to provocate a loss of their financial autonomy. A large number of painful patients thus find themselves in situations of social vulnerability even of precariousness often denied and difficult to detect by the caring team. Precarity is define as " the lack of one or several securities, in particular the employment, allowing the people and the families to assume their professional, family or social obligations, and to enjoy their fundamental rights." To allow a earlier identification of the populations in deprivation situation, the questionnaire EPICES (Evaluation of the Precariousness and the Disparities of health for the Centers of Examination of Health (CES)) was administered to more than 7000 people. The individual score, indicator of the precariousness and the disparities of health, is calculated after answer to 11 questions and was calculated on about 200 000 French people. Among numerous indicators, it appears that the consumption of psychotropics or a negative perception of the health are socioeconomic indicators, mode of life and health which are prevailing according to the quintiles of the score EPICES.

This national study, on the French CETD aims is: 1 - to study prevalence of the social vulnerability even of the precariousness thanks to adapted questionnaires of which the questionnaire EPICES, 2 - to identify predictive social-economic factors which generate and amplify this circumstance, 3 - to identify the patients for whom a situation of precariousness and social vulnerability is proved true, justifying the earlier orientation towards the social worker of the Center so allowing a "global" care of the patient during the second visit

DETAILED DESCRIPTION:
This national study is the first study on the chronic pain and the social vulnerability, as well at the level national as international because at this day there is no international publication dealing with this problem which begins to emerge in the structures setting in charge of the patients suffering of chronic pain. A recent article (Denk and al, on 2014) underlines the importance to look for the predictive factors of the chronic pain. This epidemiological study of prevalence of the social vulnerability even of the precariousness as well as predictive factors of this circumstance will allow to identify the patients with risk in a earlier way and to refer them as soon as possible for a support in the social domain. In a completely empirical way we notice important obstacles of psychosocial and societal order during the therapeutic care of the patients. This study will allow to bring important information on a troop about one thousand patients distributed on the French CETD.

ELIGIBILITY:
Inclusion Criteria:

* Patient follow-up in a CETD, Patient of more than 18 years old, Patient having a sufficient cooperation and an understanding to conform to the imperatives of the study, Patient agreeing to give a written consent, Patient member in the social security system French.

Exclusion Criteria:

* Old Patient under age 18, Patient with cooperation and understanding not allowing conforming in a strict way to the conditions and to the tests planned by the protocol, Patient benefiting from a legal protective measure (guardianship, supervision) Unaffiliated patient in the social security system French

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients follow-up in a CETD
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Estimate prevalence of the precariousness and the disparities of health at the chronic painful patient in CETD by the questionnaire EPICES | At day 1
  Estimate prevalence of the precariousness and the disparities of health at the chronic painful patient in CETD by the questionnaire EPICES (Evaluation of the Precariousness and the Disparities of Health for the Centers of Examination of Health).
  Patient which have a score EPICES ≥ 30, 2. will be considered as " vulnerable socially or precarious" and will came for a second consultation in the center of Evaluation and Treatment of the Pain, to benefit an earlier orientation and better adapted with a social worker.

SECONDARY OUTCOMES:
Estimation of the relation between precariousness / disparities of health and the quality of life estimated by the SF36 | At day 1

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France